#### **Study Protocol**

# **Official Title:**

# Comparison of Complication Rates of Onlay vs Sublay Mesh Repair of Incisional Hernia Brief Title:

Complication Rate of Onlay vs Sublay Mesh Repair in Incisional Hernia

# ClinicalTrials.gov Identifier:

NCT ID: Not Yet Assigned

# **Organization's Unique Protocol ID:**

HMC-QAD-F No. IREB-1221

## **Study Type:**

Interventional Study (Randomized Controlled Trial)

#### **Study Design:**

Parallel Assignment, Open Label

# **Sponsor:**

Hayatabad Medical Complex, Peshawar, Pakistan

# **Responsible Party:**

Principal Investigator

#### **Principal Investigator:**

Dr. Gohar Ali

Principal Investigator

Department of Surgery

Hayatabad Medical Complex, Peshawar, Pakistan

#### **Ethics Approval:**

Approved by Ethical Committee, Hayatabad Medical Complex, Peshawar

Approval Number: HMC-QAD-F No. IREB-1221

#### **Study Start Date:**

01 August 2020

#### **Primary Completion Date:**

31 August 2025

#### **Study Completion Date:**

15 September 2025

Study Design: Open-label, parallel group, randomized controlled trial

#### **Objective:**

To compare postoperative complication rates between **onlay** and **sublay** mesh repair in adult patients with incisional hernia.

## **Study Population:**

- Inclusion Criteria:
  - o Adults aged 18–60 years
  - o Primary incisional hernia
  - o Fit for open mesh repair
  - o Able to provide informed consent
- Exclusion Criteria:
  - Obstructed/strangulated hernia
  - o Recurrent hernia
  - $\circ$  BMI > 40
  - $\circ$  ASA  $\geq$  3 or severe comorbidities
  - o Unable/unwilling to follow up

Sample Size: 350

#### **Randomization:**

- Randomized 1:1 to **onlay** or **sublay** repair
- Computer-generated random sequence

#### **Interventions:**

- Experimental: Sublay Mesh Repair mesh placed in retromuscular/preperitoneal plane
- Active Comparator: Onlay Mesh Repair mesh placed over anterior rectus sheath

# **Primary Outcome:**

Postoperative complication rate within 30 days (wound infection, seroma, hematoma, recurrence)

# **Secondary Outcomes:**

- Hernia recurrence at 6 and 12 months
- Length of hospital stay
- Operative time

#### Follow-up:

• Clinical assessment on day 7, day 30, 6 months, and 12 months postoperatively

# **Ethics:**

- Approved by Institutional Review Board, HMC (HMC-QAD-F No. IREB-1221)
- Written informed consent obtained from all participants

# **Data Management:**

- Data recorded in secured database and standardized proforma
- Patient identifiers removed for any shared datasets.
- SPSS V23. Is used for data entry.